CLINICAL TRIAL: NCT05154747
Title: Long-Acting Treatment in Adolescents (LATA): A Randomised Open-label 2-arm 96 Week Trial in Virologically Suppressed HIV-1-positive Adolescents Aged 12-19 Years of Age in Sub-Saharan Africa
Brief Title: Long-Acting Treatment in Adolescents (LATA)
Acronym: LATA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Janssen-Cilag Ltd. (Industry); ViiV Healthcare (Industry); Department of Clinical Pharmacy, University Medical Centre St Radboud, The Netherlands. (Other); London School of Hygiene and Tropical Medicine (Other); MRC/UVRI and LSHTM Uganda Research Unit (Other); Africa Health Research Institute (Other); PENTA Foundation (Network); University of York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 129628
Record Dates: First submitted 2021-11-12; First posted 2021-12-13 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Hiv; HIV Infections; HIV-1-infection; Paediatric Human Immunodeficiency Virus Infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — cabotegravir, rilpivirine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous Therapy (CT) Control Group (Active Comparator): The control group is a continuous daily oral combination ART consisting of dolutegravir (DTG), with a tenofovir (TFV) and lamivudine(3TC)/emtricitabine(FTC) backbone
  Interventions: Drug: TLD
- Long Acting (LA) Injectable Group (Experimental): The intervention group is a long-acting injectable, cabotegravir (CAB) LA and rilpivirine (RPV) LA given every 8-weeks after an optional 4-week oral lead-in period with oral cabotegravir and rilpivirine, and two loading doses separated by 4 weeks.
  Interventions: Drug: Cabotegravir, Rilpivirine Drug Combination

INTERVENTIONS:
Drug: Cabotegravir, Rilpivirine Drug Combination — Cabotegravir LA 600mg as a 3mL IM injection. The product is packaged in a 3mL USP Type I glass vial. Each vial is for single-dose use. CAB LA injectable suspension is to be stored according to the product label at room temperature (<30oC). CAB LA is composed of cabotegravir free acid, polysorbate 20, polyethylene glycol3350, mannitol, and water for injection.
  Rilpivirine LA 900mg as a 3mL IM injection. Each single-dose vial contains 900mg/3mL rilpivirine. RPV LA injectable suspension should be stored according to the product label refrigerated at 2-8oC and should be protected from light. RPV LA is composed of RPV free base, poloxamer 338, sodium dihydrogen phosphate monohydrate, citric acid monohydrate, glucose monohydrate, sodium hydroxide, and water for injection.
  Cabotegravir Long-Acting (CAB LA) will be given IM into one buttock, and Rilpivirine Long-Acting (RPV LA) will be given IM into the opposite buttock.
  Other Names: CAB; RPV
  Arms: Long Acting (LA) Injectable Group
Drug: TLD — Dolutegravir 50mg oral with tenofovir disoproxil fumarate (245mg) and lamivudine (300mg) in a fixed dose combination or Dolutegravir 50mg oral with tenofovir alafenamide fumarate (25mg) and lamivudine (300mg) (l/TAF) oral in a fixed dose combination
  Arms: Continuous Therapy (CT) Control Group

SUMMARY:
The LATA trial will find out if taking a long-acting injectable form of HIV medicines, called cabotegravir and rilpivirine, every 2 month works as well as taking tablet HIV medicines every day in young people aged 12-19 years of age.

The trial is organised by an international group of researchers from Europe and Africa, and will include 460 young people, from Kenya, South Africa, Uganda and Zimbabwe.

DETAILED DESCRIPTION:
The goal of HIV treatment is to make sure the HIV virus in the blood remains very low; this is called having an undetectable viral load (virological suppression). If this goal is achieved and sustained life-long, then people with HIV infection can live a healthy life, with a normal life expectancy. However, it is challenging to take medication every single day for life. This may be an even bigger challenge for teenagers living with HIV.

There is now a new way of taking HIV treatment. This is through an injection form of the HIV medicines. Two injections, one of cabotegravir and one of rilpivirine, have to be given in the clinic every 8 weeks. One injection will be given in the left cheek of the buttock and the other in the right cheek of the buttock at the same visit. This is called an intramuscular (IM) injection.

In LATA, two different ways of taking HIV medicines will be compared. Participants will be randomised, with an equal chance that they will either go into the long-acting injectable group or get a daily tablet by mouth. This is what happens depending on which group they are randomised to:

* Long-Acting Injectable Group: In this group, there are 2 options. The first is to stay on current HIV medicines by mouth and then to start the injections around 4 weeks after randomisation. If this is the choice, then at week 4, the first 2 injections will be given, the second two will be given 4 weeks later, and then it's every 8 weeks from then on. The second option is to switch to taking one tablet of cabotegravir and one tablet of rilpivirine for approximately 4-5 weeks before starting the injections. The reason that some people might choose to have the tablet forms first, is to make sure they tolerate them. This is called an oral lead-in (OLI). For the OLI group, and as long as liver test results at 4 weeks are within normal levels, the first two injections will be given at around 5 weeks (about a week after the week 4 visit), the second two are given 4 weeks later, and then it's every 8 weeks from then on.
* Continuous Oral Treatment Group: this group will continue to take HIV medicines every day by mouth. However, to join the trial, some participants will have to change some of their oral medications as the combination being used is dolutegravir with tenofovir plus either lamivudine or emtricitabine as a single tablet taken once a day, called TLD.

The LATA trial will enrol 460 young people living with HIV-1 from Kenya, South Africa, Uganda and Zimbabwe. People taking part need to be 12 to 19 years old, HIV-1-positive, have undetectable HIV-1 viral load (HIV-1 RNA < 50 c/mL) for at least the last year, on combination ART, and never have switched HIV medication in the past because of treatment failure. In order to join, adolescents who are at least 18 years old will need to sign the consent form for themselves. The consent form describes what the trial is about and what is required of participants. Adolescents aged 12 to 17 years of age will have to sign an assent form - this assent form describes what the trial is about and what is required of participants. The assent form can be signed without a parent or guardian in the same room. The assent form has the same information in it as the consent form that their parent or guardian will also need to sign as well, to agree to them taking part in LATA. Each person taking part will stay in the trial for at least 96 weeks (about 2 years) although it may be longer, between 3-4 years. Young women enrolled in LATA must not be pregnant or breastfeeding when they join and must avoid getting pregnant during their time in the trial. For young women in the long-acting injectables group, they must also avoid getting pregnant for at least 12 months after the last injection is given; this is because not much is known about the safety of these injections in pregnancy. If, however, a young woman does get pregnant while they are on the long-acting injectables, they should immediately contact their clinic for advice and support. More details will be provided in a separate information sheet and consent form about options for HIV treatment during pregnancy, including staying on the long-acting injectables with additional monitoring.

At the beginning of the trial everyone will be screened to make sure they meet the criteria to participate, then they will be randomised - by a computer- to one of the groups in the study. For the long-acting injectable group, there are the 2 options as described above and one or two additional visits around 4-5 weeks after being randomised into the trial. People taking part in the trial will be asked to visit the clinic every 8 weeks until the last participant who joined the trial has been in the trial for 96 weeks. The trial research team will ask questions about health, wellbeing and mood at some of the visits. For girls who have started their periods, a pregnancy test will be done at each visit. Everyone will have their viral load measured approximately every 6 months and they and their doctors will receive the results, which show how much HIV virus is in the blood. At some visits a blood sample will be stored, which may be looked at later for HIV viral load or for changes to the virus that may stop some treatment working as well. An additional blood sample will also be taken at the beginning and then once a year, and urine samples at the beginning and at week 96; these stored samples will be used to look at the health of people's kidneys, bone, heart and other organ systems; they are optional. In addition, to the main trial, there are sub-studies (smaller studies within the main trial), which people taking part may be invited to take part in. Some participants in LATA will be invited to take part in a social science sub-study where there are interviews to find out how people feel about HIV and their medication. In another sub-study, the mood (neuropsychiatric) sub-study, there are additional surveys to find out if young people are having problems with feeling down or worried about HIV, their medication and other things going on in their lives. A small number of participants may be asked to take part in a study that measures the amount of HIV medicine in the blood. These sub-studies require additional consent, so people can decide if they do or don't want to take part in these sub-studies, and it won't affect being in the LATA trial. At selected sites, a further sub-study is about checking the amount of muscle and fat in the body, using a monitor placed on the arm, which doesn't hurt at all. The information for this sub-study is in the main LATA information sheet.

The trial will be able to show whether the injection forms of HIV medicine work as well as taking the daily tablets of HIV medicines in adolescents living with HIV. If the long-acting injectables given every 8 weeks work as well as the daily oral tablet, it is hoped the HIV guidelines will change to recommend this as an option for how adolescents and young people take their HIV medicines.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1-infected
2. Aged 12-19 years
3. Aware of HIV status
4. Body weight ≥35Kg
5. On ART consisting of 2NRTI and a third agent
6. On ART for ≥1 year with no previous regimen change for treatment failure*
7. Virologically suppressed with all HIV-1 RNA viral loads <50copies/mL¥ in the last 12 months up to and including screening. Additionally, there must be one result <50copies/mL at least 12 months prior to screening and the viral load at trial screening must be <50 copies/mL
8. Written informed consent provided by participant (if aged 18 to 19 years) and/or carer/legal guardian (if participant aged 12 to 17 years) as appropriate
9. Written informed assent in participants aged 12 to 17 years
10. Females who are sexually active must be willing to adhere to highly effective methods of contraception⌂

    * Treatment failure includes virological, immunological or clinical failure where regimen has been changed for lack of response to treatment

      * The screening sample VL must be <50 copies/mL. For samples prior to screening, a diluted sample may be used; if the viral load in the diluted sample is below lower limit of quantification (LLQ), a calculated VL<100 copies/mL is allowed; if the viral load in the diluted sample is equal or above LLQ the calculated VL should be below 50 copies/mL.

        * Highly effective contraception are injectable, implantable, oral and intrauterine contraceptives which have an expected failure rate <1% per year; in the LA group, must avoid pregnancy for 12 months after the last dose of the CAB and RPV LA

Exclusion Criteria:

1. Known HIV-2 infection
2. Females who are pregnant or breastfeeding
3. Females who plan to become pregnant during the trial follow-up or are sexually active and are unwilling to avoid pregnancy for the duration of the trial
4. Moderate or high-risk score on the Columbia-Suicide Severity Rating Scale
5. Hepatitis B SAg positive
6. ALT ≥3 x upper limit of normal
7. On treatment for active TB
8. Known contraindication to receipt of dolutegravir, cabotegravir, rilpivirine, emtricitabine/ lamivudine and any formulation of tenofovir
9. Participants determined by the investigator to have a high risk of seizure, including those with unstable or poorly controlled seizure disorder
10. Unwilling or contraindication to receiving injections
11. Contraindication to receiving injectable agents in the buttock area
12. Underlying medical condition (e.g. bleeding disorder; use of warfarin) that in the opinion of the investigator precludes participation
13. Previous randomisation in the BREATHER Plus trial
14. Known major^ resistance to non-nucleoside reverse transcriptase inhibitors or integrase inhibitors

    * Major NNRTI and INSTI mutations are those listed in the IAS report (www.iasusa.org/resources/hiv-drug-resistance-mutations/ - which is likely to change over time

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 476 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Confirmed virological rebound | Up to 96 week assessment
  The proportion of participants with confirmed virological rebound, defined as 2 consecutive plasma HIV-RNA ≥50 copies/mL at any time up to the 96 week assessment

SECONDARY OUTCOMES:
Efficacy Outcome: Proportions of participants with HIV-RNA ≥50 copies/mL | At week 48 and week 96 visits
  Proportions of participants with HIV-RNA ≥50 copies/mL at 48 and 96 weeks using a modified FDA snapshot algorithm
Efficacy Outcome: The proportion of participants with confirmed HIV-RNA ≥1000 copies/mL | Up to week 96 assessment
  The proportion of participants with HIV-RNA ≥1000 copies/mL (confirmed) by week 96
Efficacy Outcome: The proportion of participants with confirmed HIV-RNA ≥200 copies/mL | Up to week 96 assessment
  The proportion of participants with HIV-RNA ≥200 copies/mL (confirmed) by week 96
Efficacy Outcome: The number of HIV reverse transcriptase mutations | Up to week 96 assessment
  The number of HIV reverse transcriptase mutations in participants with confirmed virological rebound
Efficacy Outcome: The number of HIV integrase mutations | Up to week 96 assessment
  The number of HIV integrase mutations in participants with confirmed virological rebound
Efficacy Outcome: HIV-RNA <50 copies/mL | At 24, 48 and 96 week assessments
  HIV-RNA <50 copies/mL at 24, 48 and 96 weeks
Safety Outcome: Change in lipids | From baseline 96 weeks
  Changes in lipids from baseline to 96 weeks
Safety Outcome: Change in HbA1c | From baseline to 96 weeks
  Changes in HbA1c from baseline to 96 weeks
Safety Outcome: Change in Phosphate | From baseline to 96 weeks
  Changes in phosphate from baseline to 96 weeks
Safety Outcome: Change in liver function: measurement of alanine aminotransferase (ALT) | From baseline to 96 weeks
  Changes in ALT from baseline to 96 weeks
Safety Outcome: Change in renal function: measurement of eGFR | From baseline to 96 weeks
  Changes in eGFR from baseline to 96 weeks
Safety Outcome: Weight changes | From baseline to 48 and 96 weeks
  Changes in weight from baseline to 48 and 96 weeks
Safety Outcome: Height changes | From baseline to 48 and 96 weeks
  Changes in height from baseline to 48 and 96 weeks
Safety Outcome: Change in resting pulse | From baseline to 48 and 96 weeks
  Changes in resting pulse from baseline to 48 and 96 weeks
Safety Outcome: Change in blood pressure | From baseline to 48 and 96 weeks
  Changes in blood pressure from baseline to 48 and 96 weeks
Safety Outcome: Time to new or recurrent WHO grade 3 or WHO grade 4 event or death | From baseline to 96 weeks
  Time to any new or recurrent WHO grade 3 or WHO grade 4 event or death
Safety Outcome: Incidence of serious, grade 3, 4 and 5, and any treatment-modifying adverse events | From baseline to 96 weeks
  Incidence of serious, grade 3, 4 and 5, and treatment-modifying (of any grade) adverse events
Safety Outcome: The proportion of participants with any change from baseline ART regimen | From baseline to 96 weeks
  The proportion of participants with any change from baseline ART regimen
Safety Outcome: Change in CD4+ and CD8+ T-cell count | From baseline to 48 and 96 weeks
  Change in CD4+ and CD8+ T-cell count from baseline to 48 and 96 weeks
Safety Outcome: incidence of injection-site reactions of any grade | From baseline to 96 weeks
  LA group only: incidence of injection-site reactions of any grade

OTHER OUTCOMES:
Patient-Reported Outcome: Adherence to trial medications questionnaire | From baseline to 96 weeks
  Patient-reported adherence to trial medications via a short series of questions (questionnaire). The questionnaire includes items on how they take medications (do they take them independently, do they need reminders, does their parent/carer give them), and have they missed any pills since the last trial visit (if yes, how many).
Patient-Reported Outcome: Acceptability and Wellbeing | From baseline to 96 weeks
  Patient-reported acceptability and wellbeing using the HIV/AIDS-targeted quality of life (HAT-QoL) questionnaire
Patient-Reported Outcome: Depression | From baseline to 96 weeks
  Patient-reported depression using the Patient Health Questionnaire-9 (PHQ-9)
Patient-Reported Outcome: Anxiety | From baseline to 96 weeks
  Patient-reported anxiety using the Generalised Anxiety Disorder Assessment (GAD-7)
Patient-Reported Outcome: Sleep Disturbance | From baseline to 96 weeks
  Patient-reported sleep disturbances from baseline to 96 weeks using a modified Pittsburgh Sleep Questionnaire. This questionnaire measures answers to a series of sleep-related questions cover topics on breathing and snoring, fatigue and tiredness. The questionnaire utilises a 5-point Likert scale where agreement with the statements posed indicates a worse outcome.
Patient-Reported Outcome: Perception of injection questionnaire | From baseline to 96 weeks
  LA group only: perception of injection (PIN) questionnaire. The PIN questionnaire explores both pain at injection site and injection site reactions (ISR), anxiety before and after injection, willingness to receive HIV injectable treatment and satisfaction with mode of treatment administration of individuals receiving injection and perceptions associated with receiving injections. This measure contains 21 items: pain at injection site, local site reactions, impact on functioning and willingness to pursue injectable treatment outside clinical trial. Scores range from 1 to 5; questions are phrased to ensure that 1:most favourable perception of injection, and 5:most unfavourable. Higher scores represent worse perception of injection
Patient-Reported Outcome: Healthcare resource utilisation | From baseline to 96 weeks
  Healthcare resource utilisation (as a sub-study outcome)
Patient-Reported Outcome: Health-related quality-of-life | From baseline to 96 weeks
  Health-related quality-of-life (as a sub-study outcome) using the EuroQol-5 Dimension (EQ-5D) questionnaire. This questionnaire includes a scale of 0-100 where a higher score means a better outcome
Patient-Reported Outcome: Perception of body shape using Stunkard figure rating scales | From baseline to 96 weeks
  Perception of body shape using Stunkard figure rating scales (as a sub-study outcome). This is a scale from 1-9 and a higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Pett, Principal Investigator — MRC CTU at University College London
Locations (5):
- Moi University, Eldoret, Kenya
- Enhancing Care Foundation King Edward VIII Hospital, Durban, South Africa
- Uganda (2):
  - Baylor College of Medicine Childrens Foundation Uganda, Kampala
  - Joint Clinical Research Centre, Kampala
- University of Zimbabwe Clinical Research Centre, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Data collected in the study will be available for additional research with justified scientific objectives. LATA will follow a controlled access approach to making data available outside of the trial whereby researchers make formal applications for data sharing. Where a proposal has been approved, the required Individual Participant Data (IPD) will be shared with the researchers on the Data Sharing Agreement to meet the requirements of the proposal. Proposals should be sent to mrcctu.lata@ucl.ac.uk. Further information on criteria and application can be found on the MRC CTU webpage on data sharing at the following link https://www.mrcctu.ucl.ac.uk/our-research/other-research-policy/data-sharing/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be made available as per agreed timelines following approval of a data sharing request (which is unlikely to be approved before the primary trial publication).
Access Criteria: There is a controlled access approach whereby access to trial data can be requested by qualified researchers engaging in independent scientific research. As per the MRC CTU at UCL's Data Sharing and Data Reuse SOP, access will be provided following a formal application detailing the specific requirements, proposed research, qualification of researchers and publication plan, and execution of a Data Sharing Agreement. For more information or to submit a request, please contact mrcctu.lata@ucl.ac.uk.

REFERENCES:
- [Derived] Anena D, Chappell E, Nazzinda R, Kiilu C, Chitsamatanga M, Arumugam T, Green A, Kityo Mutuluuza C, Bwakura-Dangarembizi M, Siika A, Archary M, Jafta L, Namukwaya S, Seeley J, Akabwai G, Mugerwa H, Bevers L, Burger D, Walker S, Bamford A, South A, Apoto N, Bush M, Thomason MJ, Spittle B, Ford D, Kekitiinwa AR, Pett SL; LATA Trial Team. Trial design and enrolment characteristics of LATA (Long-Acting Treatment in Adolescents): A randomised, open-label, non-inferiority, 96-week trial evaluating the virological efficacy, safety, acceptability and quality-of-life of the dual long-acting injectable regimen cabotegravir/ rilpivirine compared to daily oral therapy in virologically suppressed adolescents with HIV-1 infection, aged 12 to <20 years, in Sub-Saharan Africa. Contemp Clin Trials. 2026 Jan 7:108213. doi: 10.1016/j.cct.2025.108213. Online ahead of print. PMID 41512916